CLINICAL TRIAL: NCT02264314
Title: Tele-educative Program to Improve Adherence to the Use of Hearing Aids in Patients With Hearing Loss: a Randomized Clinical Trial
Brief Title: Tele-educative Program to Improve Adherence to the Use of Hearing Aids in Patients With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Principal Investigator, Felipe Cardemil, MD, University of Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UChile
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Hearing Loss
Keywords: Aged; Hearing Aids; Rehabilitation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): This group received an audiological rehabilitation program with a tele-educative intervention boost
  Interventions: Behavioral: Active Communication Education Program
- Control (Placebo Comparator): This group received no intervention
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Active Communication Education Program — A behavioral intervention aimed to improve the adherence to the hearing aid in older adults with hearing loss
  Other Names: ACE Program
  Arms: Intervention
Other: Control — Participants in this arm will not receive intervention during the study protocol time. After the completion of the protocol, they will receive the same intervention that the intervention group, meaning the ACE program intervention.
  Other Names: Regular assistance
  Arms: Control

SUMMARY:
Hearing loss is the third most common chronic condition in over 65 years people, it is estimated that 77.8% of older adults suffer from it. However, there are reports of adherence to the use of hearing aids of only to 40%. The objective of this project is to measure the effectiveness of a tele-educative intervention to improve adherence to the use of hearing aids. A randomized controlled trial was performed. The active branch consists of the implementation of an educational program called Active Communication Education, consisting of 4 sessions with a trained rehabilitator. Participants will be also monitored by telephone headset use by personnel trained for three months. The control arm will consist of the usual care received by these patients. All participants will be assessed at home at 3, 6, 9, and 12 months after randomization.

DETAILED DESCRIPTION:
Introduction: Hearing loss is the third most common chronic condition in over 65 years people, it is estimated that 77.8% of older adults suffer from it. Delivery of hearing aids to older adults with bilateral hearing loss is included in the Garantías Explícitas en Salud (GES) Guidelines of Chile. However, there are reports of adherence to the use of hearing aids of only to 40%. The GES guideline establishes the conducting of programs in audiological rehabilitation counseling, but there is no evidence that this is being developed in Chile.

Objective: The objective of this project is to measure the effectiveness of a tele-educative intervention to improve adherence to the use of hearing aids.

Material and Methods: A randomized controlled trial was performed. Demographic and audiometric variables were recorded. The active branch consists of the implementation of an educational program called Active Communication Education, consisting of 4 sessions with a trained rehabilitator. Participants will be also monitored by telephone headset use by personnel trained for three months. The control arm will consist of the usual care received by these patients. All participants will be assessed at home at 3, 6, 9, and 12 months after randomization. The primary outcome will assess adherence to the use of hearing aids. Secondarily related quality of life was assessed with hearing loss.

Analysis Plan: Data will be analyzed mediantes bivariate tests, student t for normally distributed continuous variables, and Fisher exact test for categorical variables. A model of multilevel mixed effects will be drawn considering the repeated measurements of outcomes assessed. For all analysis is considered an alpha=5%.

ELIGIBILITY:
Inclusion Criteria:

* Hearing loss worst than 40 db in the better ear
* 65 years old or more

Exclusion Criteria:

* Dementia
* Prior surgery for hearing loss

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adherence to the hearing aid | at 12 months

SECONDARY OUTCOMES:
Quality of life | at 12 months